CLINICAL TRIAL: NCT04680598
Title: Comparison of Hepatitis B Virus Reactivation Between Patients With High HBV-DNA and Low HBV-DNA Loads Undergoing Immune Checkpoint Inhibitor and Concurrent Antiviral Prophylaxis: a Prospective Observational Study
Brief Title: Comparison of HBV Reactivation Between Patients With High HBV-DNA and Low HBV-DNA Loads Undergoing ICI and Concurrent Antiviral Prophylaxis: a Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Kaiping Central Hospital (Other); Guangzhou No.12 People's Hospital (Other Government); ZhongShan People 's Hospital (Unknown)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Other Study IDs: SH003
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high HBV-DNA group: patients with HBV-DNA >500 IU/ml
  Interventions: Drug: ICI; Drug: Antiviral Prophylaxis
- low HBV-DNA group: patients with HBV-DNA≤500 IU/ml
  Interventions: Drug: ICI; Drug: Antiviral Prophylaxis

INTERVENTIONS:
Drug: ICI — Patients received ICI, including PD-1 inhibitor (pembrolizumab, toripalimab, nivolumab, sintilimab, camrelizumab) or PD-L1 inhibitor (atezolizumab)
Drug: Antiviral Prophylaxis — Patient received concurrent antiviral prophylaxis, such as tenofovir, entecavir

SUMMARY:
Immune checkpoint inhibitor (ICI), including programmed cell death protein-1 (PD-1) inhibitor or programmed cell death-Ligand 1 (PD-L1) inhibitor , is recommended to treat advanced hepatocellular carcinoma (HCC). However, the safety of ICI in patients with a high HBV-DNA load is unknown because of the potential risk of hepatitis B virus (HBV) reactivation. This study was to compare the HBV reactivation between patients with low HBV-DNA loads and high HBV-DNA loads undergoing antiviral prophylaxis and ICI.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Seropositive for hepatitis B surface antigen (HBsAg)
* Received concurrent antiviral prophylaxis and at least one cycle of ICI treatment. Prior use of antiviral therapy was allowed
* Adherence to antiviral therapy
* A life expectancy of 3 months or more
* An Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2

Exclusion Criteria:

* other positive viral markers, including IgM antibodies to hepatitis A virus, the hepatitis C virus viral load, IgG antibodies to hepatitis D virus, IgM antibodies to hepatitis E virus
* Antibodies to human immunodeficiency virus,
* A lack of HBV DNA and liver function testing before the first immunotherapy and during the follow-up period.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible patients were divided into low HBV-DNA group (low group, ≤500 IU/ml) and high HBV-DNA group (high group, >500 IU/ml) according to baseline HBV-DNA level. Baseline HBV-DNA was the HBV-DNA level within 2 weeks prior to initial ICI therapy. For patients who had prior experience with antiviral therapy, the antiviral therapy would be continued. For patients who did not have prior experience with antiviral therapy, antiviral therapy would be administered after patients was confirmed with positive HBsAg or positive HBV-DNA level. Prior use of antiviral therapy was defined that patients have taken antiviral therapy for a period of time before they received ICI therapy. Antiviral prophylaxis was defined as anti-HBV treatment administered before and during ICI therapy. Antiviral treatment was continued even though ICI therapy was terminated.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-12-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
HBV Reactivation rate | 2 months
  HBV Reactivation rate was defined as one of the following according to the American Association for the Study of Liver Diseases (AASLD) 2018 hepatitis B guidelines: (i) a ≥2 log (100-fold) increase in HBV DNA compared to the baseline level, (ii) HBV DNA ≥3 log (1,000) IU/mL in a patient with previously undetectable level (since HBV DNA levels fluctuate)

SECONDARY OUTCOMES:
HBV-associated hepatitis | 2 months
  HBV-associated hepatitis was defined as HBV Reactivation plus an ALT increase to ≥3 times the baseline level and >100 U/L according to the AASLD 2018 Hepatitis B Guidance
PD-1 inhibitor disruption due to hepatitis | 2 months
  PD-1 inhibitor disruption due to hepatitis was defined as either premature termination or a delay of at least 7 days between PD-1 inhibitor cycles because of hepatitis.
overall survival | 12 months
adverse event | 30 Days after ICI

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospital, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong
  - ZhongShan People 's Hospital, Zhongshan